CLINICAL TRIAL: NCT05537376
Title: A Novel Peer-Delivered Recovery-Focused Suicide Prevention Intervention for Veterans With Serious Mental Illness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D4239-W
Record Dates: First submitted 2022-09-07; First posted 2022-09-13 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Psychotic Disorders; Bipolar Disorders; Suicidal Ideation; Suicide, Attempted
MeSH Terms: conditions — Psychotic Disorders; Bipolar Disorder; Suicidal Ideation; Suicide, Attempted | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: Veterans receiving SUPPORT will be offered all modules of the intervention via weekly, 50-minute sessions with a Peer Specialist. Following the completion of a mental health evaluation by a licensed professional, the Peer Specialist leads the Veteran who is at risk for suicide through recovery planning that is tailored to the Veteran's suicidal experiences with cognitive learning strategies to enhance recall of the Veteran's safety plan and improve recovery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SUPPORT (Experimental): Veterans receiving SUPPORT will be offered all modules of the intervention via weekly, 50-minute sessions with a Peer Specialist. Following the completion of a mental health evaluation by a licensed professional, the Peer Specialist leads the Veteran who is at risk for suicide through recovery planning that is tailored to the Veteran's suicidal experiences with cognitive learning strategies to enhance recall of the Veteran's safety plan and improve recovery.
  Interventions: Behavioral: SUicide Prevention by Peers Offering Recovery Tactics
- ESC (No Intervention): The enhanced standard care (ESC) condition contains the elements of standard practice suicide prevention delivered at VHA, which include: 1) suicide risk assessment, 2) VA Safety Planning Intervention, 3) timely referral to VA mental health outpatient care, and 4) Suicide Prevention Coordinator follow-up contacts. It is enhanced due to the contact with the research study.

INTERVENTIONS:
Behavioral: SUicide Prevention by Peers Offering Recovery Tactics — Following the completion of a comprehensive mental health evaluation by a licensed VA provider, which includes a suicide safety plan, if a Veteran is having active thoughts of suicide or made a suicide attempt in past three months, they may be eligible for SUPPORT. In SUPPORT, the Peer Specialist and Veteran co-create a personalized suicide-focused recovery plan (SUPPORT Plan) in flexible, 50-minute weekly encounters. The SUPPORT Plan includes modules that focus on valuing recovery, building a hope kit and daily plan, setting recovery goals, and looking ahead to enhance the Veteran's safety plan. Learning strategies are incorporated into each module to promote salience and recall of intervention material. The Peer Specialist works closely with the Veteran's treatment team and uses the most recent safety plan in the Veteran's chart to help complete the SUPPORT Plan as well as reinforce the usage of the Veteran's safety plan.
  Other Names: SUPPORT
  Arms: SUPPORT

SUMMARY:
Suicide is a major public health concern, particularly among Veterans with serious mental illness (SMI, i.e., psychotic disorders or bipolar disorders). Wellness Recovery Action Plan (WRAP) is a well-established evidence-based practice for those with SMI that centers on identifying warning signs of mental illness, developing wellness tools for functional independence, planning for day-to-day effective living within one's community, and building an action plan to create a valued life worth living. This proposed study will refine and pilot SUicide Prevention by Peers Offering Recovery Tactics (SUPPORT), a novel integrated recovery program that is an adaptation of peer-delivered WRAP for Veterans with SMI. In SUPPORT, a Peer Specialist leads a Veteran at increased risk for suicide through recovery planning that is tailored to the Veteran's suicidal experiences with cognitive learning strategies to enhance safety plan recall and improve functioning.

DETAILED DESCRIPTION:
This 5-year study aims to refine and pilot a peer-delivered intervention to improve functional and social recovery to decrease suicide risk; the study consists of two phases. Phase 1 employs a user-centered design approach to refine SUicide Prevention by Peers Offering Recovery Tactics (SUPPORT) aided by scientific and consumer advisory board stakeholders as well as training Peer Specialists to fidelity on pilot cases in an open trial. SUPPORT is a flexibly delivered intervention intended to augment safety planning by addressing functional and social goals personalized to each Veteran's recovery following a suicidal crisis while including cognitive learning strategies to enhance recall and salience of intervention material. Following adaptations from Phase 1, Phase 2 includes a pilot randomized controlled trial of SUPPORT compared to an enhanced standard care condition. Veteran participants in both phases will be quantitatively assessed at baseline, mid-treatment, post-treatment, and 3-months post-treatment (and qualitatively interviewed at post-treatment). Peer Specialists delivering the intervention will also be qualitatively interviewed post-treatment. The primary outcomes to be evaluated is improvement in personal recovery and reduction in suicidal ideation severity. Secondary outcomes concern changes in various domains of personal and social functioning.

ELIGIBILITY:
Inclusion Criteria:

Veteran Inclusion Criteria:

1. Veterans who report present suicidal ideation (i.e., Columbia-Suicide Severity Rating Scale (C-SSRS) > 2 ("Active thoughts of killing oneself") in past 1 month and/or a suicide attempt in the prior 3 months as identified by the C-SSRS
2. Current SMI diagnosis (i.e., schizophrenia and other psychotic disorders, mood disorders with psychotic features, bipolar disorders)
3. Capable of informed consent via the University of California San Diego Brief Assessment of Capacity to Consent (UBACC)

Peer Specialist Inclusion Criteria:

1. Certified Peer Specialist employed at VA San Diego Healthcare System (VASDHS) in the Mental Health Care Line (individuals must demonstrate competency in basic suicide screening and referral procedures to be certified)
2. 2-3 years of experience post certification as a Certified Peer Specialist
3. Interest in being trained in SUPPORT
4. Provide verbal or written consent for the research staff to discuss ability to participate in the study with the Peer Specialist's direct clinical supervisor
5. Direct clinical supervisor agreement to allow the Peer Specialist to participate. This includes the Peer Specialist's direct clinical supervisor agreement to allow the Peer Specialist time as part of their current scope of practice to 1) participate in the full day (8-hour) SUPPORT training, 2) participate in weekly 1-hour group supervision for the duration of the Peer Specialist's time in the study, and 3) take on a case load of at least one SUPPORT Veteran at a given time.

Exclusion Criteria:

Veteran Exclusion Criteria:

1. Cannot complete the assessment battery
2. Current intoxication requiring immediate detoxification or outpatient plan directed specifically to residential substance use disorder (not mental health) services
3. Imminent psychiatric hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2023-09-12 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of recruitment and retention | Through study completion, an average of 4 years
  Recruitment and retention is determined by the number of participants who were initially contacted, consented, completed baseline data, and completed follow-up data.
Acceptability of SUPPORT as measured by the Client Satisfaction Questionniare-8 (CSQ-8) | At the end of the intervention, an average of 4-weeks
  The CSQ-8 brief survey has been used extensively in VA and non-VA settings to assess overall satisfaction with care, and it has excellent internal consistency (0.93). An overall score" is calculated by summing the participant's rating score for each scale item. Scores range from 8 to 32, with higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
Change in the Scale for Suicide Ideation (SSI) | Baseline, 2-weeks, 4-weeks, 3-month follow-up
  The SSI is an 19-item interviewer administered assessment of suicidal ideation (SI) severity. The total score ranges from 0 to 38 with higher scores indicating more serve SI. The scale has demonstrated strong validity and reliability.
Change in Recovery Assessment Scale-41 | Baseline, 2-weeks, 4-weeks, 3-month follow-up
  The RAS-41 is a self-report measure of personal recovery with five domains: personal confidence and hope; willingness to ask for help; goal and success orientation; reliance on others; no domination by symptoms. A review study found high Cronbach's alphas (.76 and .97) and test-retest reliability (.65 to .88). The RAS has been widely used in VA and non-VA clinical trial studies with diverse populations, a range of mental illnesses, and has demonstrated sensitivity to change over time.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha A Chalker, PhD, Principal Investigator — VA San Diego Healthcare System, San Diego, CA
Locations (1):
- VA San Diego Healthcare System, San Diego, CA, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chalker S, Carter J, Imai Y, Depp C, Chinman M. A Recovery-Oriented Suicide Prevention Program Led by Peer Specialists for Veterans With Serious Mental Illness: Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2025 Aug 20;14:e66182. doi: 10.2196/66182. PMID 40834400
- [Derived] Chalker SA, Serafez J, Imai Y, Stinchcomb J, Mendez E, Depp CA, Twamley EW, Fortuna KL, Goodman M, Chinman M. Suicide Prevention by Peers Offering Recovery Tactics (SUPPORT) for US Veterans With Serious Mental Illness: Community Engagement Approach. J Particip Med. 2024 May 23;16:e56204. doi: 10.2196/56204. PMID 38781010